CLINICAL TRIAL: NCT01834534
Title: Telemonitoring Enhanced Support for Depression Self Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James Aikens, PhD, Associate Professor of Family Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MH096699 (NIH); 1R01MH096699-01 (NIH)
Record Dates: First submitted 2012-09-13; First posted 2013-04-18 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CarePartners for depression (Experimental): For one year, patients receive weekly automated telemonitoring of mood and self-management, while their CarePartners receive weekly reports of the patient's assessment results with tailored instructions on supporting the patient's depression self-management.
  Interventions: Behavioral: CarePartners for depression
- Usual care (No Intervention): Usual medical care.

INTERVENTIONS:
Behavioral: CarePartners for depression — Automated telephone calls for depression monitoring and self-management support.
  Arms: CarePartners for depression

SUMMARY:
The objective of this research is to test the efficacy of "CarePartners for Depression" (CP-D) intervention, which was designed to increase between visit monitoring of depression status and enhance self-management.

**In order to participate, subjects must be patients at participating clinics: Alcona Health Center, Cherry Street Health Services, Dua Family Practice, Morang Chester.

DETAILED DESCRIPTION:
This project will test a practical intervention that uses low cost technologies to activate depressed patients' existing social networks for self-management support. The intervention links patients with a "CarePartner" (CP), i.e., a non-household family member or close friend who is willing to support the patient in coordination with the clinician and any existing in-home caregiver (ICG). Through weekly automated telemonitoring, patients report their mood and self-management status, and receive tailored guidance on self-management. The CP receives a corresponding update along with guidance on how to best support the patient's self-management efforts, and the primary care team is notified about clinically urgent situations. The intervention will be tested among depressed primary care patients from clinics serving low-income and underinsured patients, whom the intervention was especially designed to benefit. Specific Aim 1 is to conduct a randomized controlled trial to compare the effectiveness of one year of telemonitoring-supported CP for depression versus usual care (control) on depression severity. Specific Aim 2 is to examine key secondary outcomes (response and remission, impairment, well-being, caregiving burden, healthcare costs) and potential moderators. Specific Aim 3 is to use a mixed-methods approach to enrich our interpretation of the statistical associations, and to discover strategies to enhance the intervention's acceptability, effectiveness, and sustainability. If the intervention proves effective without increasing clinician burden or marginal costs, then its subsequent implementation could yield major public health benefits, especially in medically underserved populations.

ELIGIBILITY:
NOTE: In order to participate, must have received medical care for past year at one of the participating clinics: Alcona Health Center, Cherry Street Health Services, Dua Family Practice, Morang Chester

Additional Inclusion Criteria:

* at least 2 outpatient primary care visits in the past 2 years, 1 within the past 13 months
* depression diagnosis in medical chart problem list or billing record (ICD9 codes: 296.20-.26, .30-.36, 296.4-.9, 298.0, 300.4, 309.0-.1, 309.28, 311.00) during the past 2 years
* current PHQ >10 (non-mild depressive symptoms)
* at least 21 years old
* comfortable speaking English
* can use a touch-tone phone
* can identify at least 1 eligible CarePartner
* not in palliative care, on transplant waitlist, or <1 year life expectancy
* free of major cognitive impairment or psychiatrically unstable
* not experiencing domestic abuse or stalking

Exclusion Criteria:

* Limited life expectancy (e.g., advanced stage cancer/heart failure/on oxygen/end stage renal disease), receiving palliative care
* At risk for domestic abuse, PHQ<10, end stage renal disease, lung cancer, dementia, bipolar disease, schizophrenia, limited life expectancy (advanced stage cancer/heart failure/on oxygen), alcohol problems, receiving palliative care
* Unable to speak English
* Not planning to get all or most of care at study site
* Primary care physician not affiliated with study site
* Unable to use telephone to respond to weekly automated self-management support calls
* Unable to nominate an eligible CP

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2013-09; Primary Completion 2018-05-29 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Depressive symptom severity | 12 months after randomization
  Patient Health Questionnaire 9 (PHQ-9).

SECONDARY OUTCOMES:
Depression remission rate | 12 months after randomization
  Remission as measured by PHQ-9 <10
Depression-related functional impairment | 12 months after randomization
  Sheehan Disability Scale
Positive well-being | 12 months after randomization
  Positive well-being will be assessed using the REMIT, a 5-item scale of positive affect and other aspects of depression recovery developed by the PI and his colleagues. Reference: Nease DE, Jr., Aikens, JE, Klinkman, MK, Kroenke, K, and Sen, A. Toward a more comprehensive assessment of depression remission: the Remission Evaluation and Mood Inventory Tool (REMIT). Journal of General Hospital Psychiatry. 2011.
Health care costs | 12 months after randomization
  Health care costs will be estimated using data gathered from a variety of patient self-report and site-specific administrative databases.

CONTACTS AND LOCATIONS:
Overall Officials: James E Aikens, Ph.D., Principal Investigator — University of Michigan; John D Piette, Ph.D., Principal Investigator — University of Michigan
Locations (7):
- United States (7):
  - Alcona Health Centers, Alpena, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Dua Family Practice, Canton, Michigan
  - Morang Chester, Detroit, Michigan
  - Hamilton Community Health Network, Inc., Flint, Michigan
  - Cherry Street Health Services, Grand Rapids, Michigan
  - Muskegon Family Care, Muskegon Heights, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Javier SJ, Risbud R, Rossi FS, Slightam C, Aikens J, Guetterman T, Piette JD, Trivedi R. Improving depression management with support from close others: A thematic analysis of individuals with depression and their partners in care. Chronic Illn. 2024 Jun;20(2):283-295. doi: 10.1177/17423953231175690. Epub 2023 Oct 30. PMID 37904531
- [Derived] Aikens JE, Valenstein M, Plegue MA, Sen A, Marinec N, Achtyes E, Piette JD. Technology-Facilitated Depression Self-Management Linked with Lay Supporters and Primary Care Clinics: Randomized Controlled Trial in a Low-Income Sample. Telemed J E Health. 2022 Mar;28(3):399-406. doi: 10.1089/tmj.2021.0042. Epub 2021 Jun 4. PMID 34086485